CLINICAL TRIAL: NCT05808972
Title: 0.9% Sodium Chloride Versus Ringer's Lactate in the Treatment of Severe Diabetic Ketoacidosis: a Randomized Trial
Brief Title: 0.9% Saline Versus Balanced Solutions in Severe Diabetic Ketoacidosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tunis University (Other)
Responsible Party: Principal Investigator, Ahlem Trifi, Associate Professor, Tunis University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Rabta-ICU
Record Dates: First submitted 2023-03-16; First posted 2023-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Metabolic Ketoacidosis; Ketoacidemia; Acetonemia; Acetonuria
Keywords: Severe diabetic ketoacidosis,; Sodium chloride 0.9%; Ringer lactate; Base excess
MeSH Terms: conditions — Ketosis; Diabetic Ketoacidosis | interventions — Sodium Chloride; Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: Independant groups included by randomisation
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sodium chloride 0.9% (SC) arm (Active Comparator): The SC arm receives insulin therapy via an electric syringe (Actrapid HM ®, Novorapide®) (1 ml = 100 IU) - take 0.5 ml (= 40 IU) and complete to 50 ml with SC to obtain a solution of 1 ml = 1 IU. -Infusion rate = 0.1 IU/kg/h.
  In parallel, and on an insulin-independent route, 0.9% chloride saline is started on the basis of 3 L/ 24 hours per day if capillary glyceamia>2,5 g/l . Blood samples were taken for glycemia, arterial Blood gas, electrolytes, lactate at baseline, 6, 12, 24 and 48 hours later.
  Interventions: Drug: Sodium chloride 0.9% (SC)
- Ringer lactate (RL) arm (Active Comparator): The SC arm receives insulin therapy via an electric syringe (Actrapid HM ®, Novorapide®) (1 ml = 100 IU) - take 0.5 ml (= 40 IU) and complete to 50 ml with SC to obtain a solution of 1 ml = 1 IU. -Infusion rate = 0.1 IU/kg/h.
  In parallel, and on an insulin-independent route, Ringer lactate is started on the basis of 3 L/ 24 hours per day if capillary glyceamia>2,5 g/l . Blood samples were taken for glycemia, arterial Blood gas, electrolytes, lactate at baseline, 6, 12, 24 and 48 hours later.
  Interventions: Drug: Ringer lactate (RL)

INTERVENTIONS:
Drug: Sodium chloride 0.9% (SC) — This trial looks specifically at the type of hydratation liquid. The patients included will receive SC. The volume, frequency of fluid administration and other severe DKA therapies, such as insulin therapy and electrolytes, are prescribed similarly. The intervention will continue for 48 hours from admission to the ICU with a blood gas control (including base excess) + Blood glucose + ionogram (Na, K, chlorine) + lactates on admission (or H0), H6, H12, H24 and H48.
  Other Names: Hydration solution
  Arms: Sodium chloride 0.9% (SC) arm
Drug: Ringer lactate (RL) — The intervention will continue for 48 hours from admission to the ICU with a blood gas control (including base excess) + Blood glucose + ionogram (Na, K, chlorine) + lactates on admission (or H0), H6, H12, H24 and H48.
  Other Names: Hydration solution
  Arms: Ringer lactate (RL) arm

SUMMARY:
Severe diabetic ketoacidosis (DKA) is a potentially serious complication of diabetes mellitus. The treatment regimen is based on insulin and rehydration. The choice of rehydration solution is a question that remains open. We sought to compare the effect of sodium chloride 0.9% (SC) versus ringer lactate (RL) in the resolution of severe DKA as well as on the variation of electrolytes.

DETAILED DESCRIPTION:
We design an open randomized trial in adult patients admitted to our ICU for severe DKA. The insulin therapy protocol was identical and the randomization concerned the rehydration solution either by SC or RL. The primary endpoint was resolution of DKA at H48 defined by a composite endpoint (glycemia <11 mmol/l, bicarbonates > 15 mmol/l or pH>7.30 and anion gap <16). The secondary endpoints were resolution of DKA at H24, change in base excess to ≥ -3 meq/L at 48 h and H24 and change in electrolytes, insulin requirements, length of stay and mortality. Blood gases, ionogram with chloride and lactate were performed at baseline, H6, H12, H24 and H48.

ELIGIBILITY:
Inclusion Criteria:

- All patients aged 16 and over hospitalized in intensive care for severe ketoacidosis defined as arterial pH ≤ 7.25 (or serum bicarbonate ≤ 15 mmol/L) and blood glucose ≥ 14 mmol/L and need for ICU.

Exclusion Criteria:

* < 16 Y

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with composite endpoint achievement | 48 hours from inclusion
  composite endpoint (glycemia <11 mmol/l, bicarbonates >15 mmol/l or pH >7.30 and anion gap <16).

SECONDARY OUTCOMES:
change in base excess to ≥ -3 meq/L | at 48 hours and at 24 hours from inclusion
  to ≥ -3 meq/L
Number of participants with hyperchloremia | at 48 hours from inclusion
  chlore level > 105 mmol/L
Total insulin dose received | through study completion, an average of 9 months
  insulin dose prescribed during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ahlem Trifi, Principal Investigator — Rabta
Locations (1):
- Ahlem Trifi, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trifi A, Ben Braik I, Galai H, Azzouz N, Tlili B, Mehdi A, Messaoud L, Seghir E, Ouhibi A, Abdellatif S. 0.9% sodium chloride versus ringer's lactate in the management of severe diabetic ketoacidosis: A randomized trial. Med Intensiva (Engl Ed). 2025 Apr 14:502203. doi: 10.1016/j.medine.2025.502203. Online ahead of print. PMID 40234173